CLINICAL TRIAL: NCT03870243
Title: Feasibility and Acceptability Followed by Effectiveness of Bubble Continuous Positive Airway Pressure (bCPAP) for Treatment of Children Aged 1-59 Months With Severe Pneumonia in Ethiopia: A Cluster Randomized Controlled Clinical Trial
Brief Title: Feasibility and Acceptability Followed by Effectiveness of bCPAP for Treatment of Children Aged 1-59 Months With Severe Pneumonia in Ethiopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Armauer Hansen Research Institute (AHRI), Ethiopia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR-18052
Record Dates: First submitted 2019-03-06; First posted 2019-03-12 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Severe Pneumonia
Keywords: Bubble CPAP; Young Children; Severe Pneumonia; Hypoxemia; Treatment failure; Mortality
MeSH Terms: conditions — Pneumonia; Hypoxia

STUDY DESIGN:
Intervention Model Description: Children aged 1-59 months with Severe Pneumonia in Ethiopia, divided in two arms; one arm will get bCPAP other arm will get WHO recommended low flow oxygen.
Masking Description: As it was an open-labeled randomized controlled clinical trial, there was no masking in any intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bubble CPAP (Active Comparator): 6 hospitals will be selected randomly for this arm
  Interventions: Device: Bubble CPAP
- Low flow oxygen (Active Comparator): 6 hospitals will be selected for low flow oxygen therapy
  Interventions: Device: Low flow oxygen

INTERVENTIONS:
Device: Bubble CPAP — To see the effectiveness of Bubble Continuous Positive Airway Pressure (bCPAP) in children with severe pneumonia
  Arms: Bubble CPAP
Device: Low flow oxygen — To see the effectiveness of low flow oxygen in children with severe pneumonia
  Arms: Low flow oxygen

SUMMARY:
Principal Investigator: Mohammod Jobayer Chisti

Research Protocol Title: Feasibility and Acceptability Followed by Effectiveness of Bubble Continuous Positive Airway Pressure (bCPAP) for Treatment of Children aged 1-59 months with Severe Pneumonia in Ethiopia: A Cluster Randomized Controlled Clinical Trial

Proposed start date: 1st July 2018, Estimated end date: 31st December 2022

Background: Feasibility and acceptability followed by effectiveness of bubble continuous positive airway pressure (CPAP) were not evaluated in childhood severe pneumonia in developing countries at a larger scale.

Objectives:

Stages I and II

* To assess the feasibility and acceptability (not only by patients' care-givers but also by physicians and nurses) of bubble CPAP in treating childhood severe pneumonia in two tertiary hospitals in Stage I and in two district hospitals in Stage II
* To record adverse events following use of bubble CPAP in these settings
* To understand how much resource and time are needed to institutionalize and maintain bubble CPAP as a routine practice in the health system

Stage III:

* To determine therapeutic efficacy/effectiveness of bubble CPAP compared to WHO standard low flow oxygen in reducing treatment failure in children admitted to hospitals with severe pneumonia and hypoxemia
* To determine therapeutic effectiveness of bubble CPAP compared to WHO standard low flow oxygen in reducing treatment failure & mortality in children aged 1-12 months admitted to hospitals with severe pneumonia and hypoxemia
* To record adverse events (pneumothorax, abdominal distension, nasal trauma, aspiration pneumonia) encountered.

DETAILED DESCRIPTION:
Methodology:

Cluster randomized controlled clinical trial

Methodology:

1. Stages I and II: Feasibility/demonstration stage will be done as an internal pilot in 3 hospitals

   a. Current treatment practice, facilities, and operational challenges will be evaluated for the introduction, clinical use and maintenance of bubble CPAP
2. Stage III: Implementation of bubble CPAP will be done in 12 hospitals a. It will be done following a cluster randomized design

Data collection-socio-demographic and clinical data will be collected using structured questionnaire by trained nurses and physicians.

Research Site:

St. Paulos Millennium Medical College, Yekatit 12 and Tikur Anbessa Specialized hospitals, 14 district hospitals

Number of Participants/Patients:

Stage I-30 children in each tertiary hospital (this stage has completed and we enrolled 49 children from two tertiary hospitals; these 49 enrolled children took double of our anticipated time {4 months}) Stage II- 20 children in each general hospital (2 general/district hospitals, we have enrolled total 40 children from this two hospitals from January 2020 to July 2020, which included COVID-19 period) Stage III-1240 children in 12 general/district hospitals (620 in bubble CPAP arm and 620 in WHO standard low flow arm; each hospital will be the cluster and 6 will be randomized to each arm)

Main Inclusion Criteria:

* Age between 1 month and 59 months
* Meet WHO clinical criteria for severe pneumonia with hypoxemia
* Hypoxemia (Oxygen saturation <90% in room air)
* Parent/guardian gives informed consent to participate in the study

Statistical Analysis:

* STATA -14: for initial two phases descriptive analysis of level of feasibility and acceptability will be performed
* For the phase III: We shall follow the principle of intention to treat. --Treatment failure and/or death will be analyzed using χ² or Fisher's exact tests as appropriate.
* Primary and secondary outcomes will be compared by calculating relative risks (RRs) and their 95% confidence intervals.
* Log-linear binomial regression will be applied to adjust for covariates to evaluate the true impact of bubble CPAP in evaluating primary and secondary outcomes and to adjust for baseline differences.
* Continuous variables will be analyzed using the Student t-test or the Mann-Whitney test as appropriate.

Study Duration:

48 months.

ELIGIBILITY:
Inclusion Criteria:

* Age between 1 month and 59 months,
* Meet WHO clinical criteria for severe pneumonia with hypoxemia.
* Oxygen saturation <90% despite standard flow oxygen therapy
* Parent/guardian gives informed consent to participate in the study

Exclusion Criteria:

* Known congenital heart disease, asthma, or upper -airway obstruction
* Tracheostomy
* Pneumothorax
* Needs mechanical ventilation for any specific reason as decided by the clinician

Ages: 1 Month to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1240 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
For stage I and II feasibility and acceptability of bubble CPAP in two tertiary and two district hospitals will be measured in number and reported in percentage | 7 months
  Patient level and health professional level challenge is the outcome of phase I and II. All will be measured in number and reported in percentage. For stage I and II: Primary outcome: operational challenges that may include availability of pulse oxymetry, IV cannula, IV antibiotics, oxygen supply system and nasal catheters for treating severe pneumonia Secondary outcomes: prevalence of severe pneumonia associated hypoxemia, their treatment practices, adverse events, mortality and treatment failure
For stage III: Primary outcome: Treatment failure | 12-18 months (Mid April 2021 to Mid October 2022)
  According to this protocol treatment failure will be declared if the following criteria are met:
  A. Presence of severe hypoxemia (SpO2<85%) at any time after at least one hour of intervention plus severe respiratory distress when the child is receiving BCPAP/LF OR, B. If the patient developed the indication of mechanical ventilation when the child is receiving BCPAP/LF OR, C. If the patient died during hospitalization OR, D. If the patient left against medical advice (LAMA) due to lack of improvement or deterioration of the child during hospitalization
  All will be measured in number and reported in percentage.

SECONDARY OUTCOMES:
Secondary outcomes: • Death • Adverse events (pneumothorax, abdominal distension, nasal trauma, aspiration pneumonia ) encountered | 12-18 months (Mid April 2021 to Mid October 2022)
  All will be measured in number and reported in percentage.

OTHER OUTCOMES:
Length of hospital stay in days | 12-18 months (Mid April 2021 to Mid October 2022)
  Length of hospital stay will be measured and reported in days.
Incidence of nasal trauma, gastric distention, shock and air leaks in number | 12-18 months (Mid April 2021 to Mid October 2022)
  Incidence of nasal trauma, gastric distention, shock and air leaks will be measured in number and reported in percentage.
Duration of bCPAP in hour | 12-18 months (Mid April 2021 to Mid October 2022)
  Duration of bCPAP will be measured and reported in hour/hours.
Acceptability of bCPAP by nurses and physicians will be measured in number and reported in percentage | 12-18 months (Mid April 2021 to Mid October 2022)
  Acceptability of bCPAP by nurses and physicians will be measured in number and reported in percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammod Jobayer Chisti, PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh (icddr,b), Dhaka, Mohakhali, Bangladesh

IPD SHARING:
Plan to Share IPD: No
We will share the final outcome after completing the study

REFERENCES:
- [Background] UNICEF. Committing to Child Survival: A Promise Renewed. Progress Report 2015 2015
- [Background] Liu L, Oza S, Hogan D, Perin J, Rudan I, Lawn JE, Cousens S, Mathers C, Black RE. Global, regional, and national causes of child mortality in 2000-13, with projections to inform post-2015 priorities: an updated systematic analysis. Lancet. 2015 Jan 31;385(9966):430-40. doi: 10.1016/S0140-6736(14)61698-6. Epub 2014 Sep 30. PMID 25280870
- [Background] You D, Hug L, Ejdemyr S, Idele P, Hogan D, Mathers C, Gerland P, New JR, Alkema L; United Nations Inter-agency Group for Child Mortality Estimation (UN IGME). Global, regional, and national levels and trends in under-5 mortality between 1990 and 2015, with scenario-based projections to 2030: a systematic analysis by the UN Inter-agency Group for Child Mortality Estimation. Lancet. 2015 Dec 5;386(10010):2275-86. doi: 10.1016/S0140-6736(15)00120-8. Epub 2015 Sep 8. PMID 26361942
- [Background] Graham SM, English M, Hazir T, Enarson P, Duke T. Challenges to improving case management of childhood pneumonia at health facilities in resource-limited settings. Bull World Health Organ. 2008 May;86(5):349-55. doi: 10.2471/blt.07.048512. PMID 18545737
- [Background] Rahman AE, Moinuddin M, Molla M, Worku A, Hurt L, Kirkwood B, Mohan SB, Mazumder S, Bhutta Z, Raza F, Mrema S, Masanja H, Kadobera D, Waiswa P, Bahl R, Zangenberg M, Muhe L; Persistent Diarrhoea Research Group. Childhood diarrhoeal deaths in seven low- and middle-income countries. Bull World Health Organ. 2014 Sep 1;92(9):664-71. doi: 10.2471/BLT.13.134809. Epub 2014 Jun 23. PMID 25378757
- [Background] Duke T, Tamburlini G, Silimperi D; Paediatric Quality Care Group. Improving the quality of paediatric care in peripheral hospitals in developing countries. Arch Dis Child. 2003 Jul;88(7):563-5. doi: 10.1136/adc.88.7.563. No abstract available. PMID 12818896
- [Background] Duke T, Peel D, Graham S, Howie S, Enarson PM, Jacobson R. Oxygen concentrators: a practical guide for clinicians and technicians in developing countries. Ann Trop Paediatr. 2010;30(2):87-101. doi: 10.1179/146532810X12637745452356. PMID 20522295
- [Background] McKiernan C, Chua LC, Visintainer PF, Allen H. High flow nasal cannulae therapy in infants with bronchiolitis. J Pediatr. 2010 Apr;156(4):634-8. doi: 10.1016/j.jpeds.2009.10.039. Epub 2009 Dec 29. PMID 20036376
- [Background] Schibler A, Pham TM, Dunster KR, Foster K, Barlow A, Gibbons K, Hough JL. Reduced intubation rates for infants after introduction of high-flow nasal prong oxygen delivery. Intensive Care Med. 2011 May;37(5):847-52. doi: 10.1007/s00134-011-2177-5. Epub 2011 Mar 3. PMID 21369809
- [Background] Duke T. CPAP: a guide for clinicians in developing countries. Paediatr Int Child Health. 2014 Feb;34(1):3-11. doi: 10.1179/2046905513Y.0000000102. Epub 2013 Dec 6. PMID 24165032
- [Background] Chisti MJ, Salam MA, Smith JH, Ahmed T, Pietroni MA, Shahunja KM, Shahid AS, Faruque AS, Ashraf H, Bardhan PK, Sharifuzzaman, Graham SM, Duke T. Bubble continuous positive airway pressure for children with severe pneumonia and hypoxaemia in Bangladesh: an open, randomised controlled trial. Lancet. 2015 Sep 12;386(9998):1057-65. doi: 10.1016/S0140-6736(15)60249-5. Epub 2015 Aug 19. PMID 26296950
- [Background] Koti J, Murki S, Gaddam P, Reddy A, Reddy MD. Bubble CPAP for respiratory distress syndrome in preterm infants. Indian Pediatr. 2010 Feb;47(2):139-43. doi: 10.1007/s13312-010-0021-6. Epub 2009 May 20. PMID 19578226
- [Background] Chisti MJ, Duke T, Ahmed T, Shahunja KM, Shahid ASMSB, G. FAS, et al. The Use of Bubble CPAP and Humidified High Flow Nasal Cannula Oxygen Therapy in Children with Severe Pneumonia and Hypoxemia: A Systematic Review of the Evidence. Bangladesh Crit Care J. 2014; 2:71-8
- [Background] Liptsen E, Aghai ZH, Pyon KH, Saslow JG, Nakhla T, Long J, Steele AM, Habib RH, Courtney SE. Work of breathing during nasal continuous positive airway pressure in preterm infants: a comparison of bubble vs variable-flow devices. J Perinatol. 2005 Jul;25(7):453-8. doi: 10.1038/sj.jp.7211325. PMID 15858606
- [Background] Courtney SE, Kahn DJ, Singh R, Habib RH. Bubble and ventilator-derived nasal continuous positive airway pressure in premature infants: work of breathing and gas exchange. J Perinatol. 2011 Jan;31(1):44-50. doi: 10.1038/jp.2010.55. Epub 2010 Apr 15. PMID 20393478
- [Background] van den Heuvel M, Blencowe H, Mittermayer K, Rylance S, Couperus A, Heikens GT, Bandsma RH. Introduction of bubble CPAP in a teaching hospital in Malawi. Ann Trop Paediatr. 2011;31(1):59-65. doi: 10.1179/1465328110Y.0000000001. PMID 21262111
- [Background] Buckmaster AG, Arnolda G, Wright IM, Foster JP, Henderson-Smart DJ. Continuous positive airway pressure therapy for infants with respiratory distress in non tertiary care centers: a randomized, controlled trial. Pediatrics. 2007 Sep;120(3):509-18. doi: 10.1542/peds.2007-0775. PMID 17766523
- [Background] Kinikar A, Kulkarni R, Valvi C, Gupte N. Use of indigenous bubble CPAP during swine flu pandemic in Pune, India. Indian J Pediatr. 2011 Oct;78(10):1216-20. doi: 10.1007/s12098-011-0389-x. Epub 2011 Mar 26. PMID 21442266
- [Background] Tagare A, Kadam S, Vaidya U, Pandit A, Patole S. A pilot study of comparison of BCPAP vs. VCPAP in preterm infants with early onset respiratory distress. J Trop Pediatr. 2010 Jun;56(3):191-4. doi: 10.1093/tropej/fmp092. Epub 2009 Oct 20. PMID 19843596
- [Background] Daga S, Mhatre S, Borhade A, Khan D. Home-made continuous positive airways pressure device may reduce mortality in neonates with respiratory distress in low-resource setting. J Trop Pediatr. 2014 Oct;60(5):343-7. doi: 10.1093/tropej/fmu023. Epub 2014 Apr 23. PMID 24760748
- [Background] Koyamaibole L, Kado J, Qovu JD, Colquhoun S, Duke T. An evaluation of bubble-CPAP in a neonatal unit in a developing country: effective respiratory support that can be applied by nurses. J Trop Pediatr. 2006 Aug;52(4):249-53. doi: 10.1093/tropej/fmi109. Epub 2005 Dec 2. PMID 16326752
- [Background] Yagui AC, Vale LA, Haddad LB, Prado C, Rossi FS, Deutsch AD, Rebello CM. Bubble CPAP versus CPAP with variable flow in newborns with respiratory distress: a randomized controlled trial. J Pediatr (Rio J). 2011 Nov-Dec;87(6):499-504. doi: 10.2223/JPED.2145. PMID 22170173
- [Background] Wilson PT, Morris MC, Biagas KV, Otupiri E, Moresky RT. A randomized clinical trial evaluating nasal continuous positive airway pressure for acute respiratory distress in a developing country. J Pediatr. 2013 May;162(5):988-92. doi: 10.1016/j.jpeds.2012.10.022. Epub 2012 Nov 16. PMID 23164308
- [Background] Federal Democratic Republic of Ethiopia Ministry of Health. Integrated Management of Newborn and Childhood Illness, Part 1 Blended Learning Module for the Health Extension Programme
- [Derived] Gebre M, Haile K, Duke T, Faruk MT, Kamal M, Kabir MF, Uddin MF, Shimelis M, Beyene T, Solomon B, Solomon M, Bayih AG, Abdissa A, Balcha TT, Argaw R, Demtse A, Weldetsadik AY, Girma A, Haile BW, Shahid ASMSB, Ahmed T, Clemens JD, Chisti MJ. Effectiveness of bubble continuous positive airway pressure for treatment of children aged 1-59 months with severe pneumonia and hypoxaemia in Ethiopia: a pragmatic cluster-randomised controlled trial. Lancet Glob Health. 2024 May;12(5):e804-e814. doi: 10.1016/S2214-109X(24)00032-9. Epub 2024 Mar 21. PMID 38522443